CLINICAL TRIAL: NCT06857513
Title: Post-ICU Syndrome Over Time in Patients With Respiratory Failure
Acronym: PICUS2
Status: Not yet recruiting | Type: Observational
Sponsor: Dr. Negrin University Hospital (Other)
Responsible Party: Principal Investigator, Ángel Becerra-Bolaños, MD PhD, Principal Investigator, Dr. Negrin University Hospital
Other Study IDs: PICUS-2025
Record Dates: First submitted 2025-02-26; First posted 2025-03-04 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Post-Intensive Care Syndrome; Quality of Life
Keywords: risk factors; intensive care unit; comorbidities
MeSH Terms: conditions — postintensive care syndrome | interventions — Physical Examination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients suffering from post-intensive care syndrome: Patients suffering from at least one symptom of post-intensive care syndrome
  Interventions: Diagnostic Test: Questionnaire and Physical Exam; Diagnostic Test: EuroQol 5-Dimension 3-Level; Diagnostic Test: EuroQol Visual Analogue Scale (EQ-VAS)
- Patients not suffering from post-intensive care syndrome: Patients without any symptom of post-intensive care syndrome
  Interventions: Diagnostic Test: Questionnaire and Physical Exam; Diagnostic Test: EuroQol 5-Dimension 3-Level; Diagnostic Test: EuroQol Visual Analogue Scale (EQ-VAS)

INTERVENTIONS:
Diagnostic Test: Questionnaire and Physical Exam — Patients will be interviewed about the current suffering of post-intensive care symptoms
Diagnostic Test: EuroQol 5-Dimension 3-Level — to assess health-related quality of life, focusing on the assessment of five key dimensions: mobility, self-care, daily activities, pain/discomfort and anxiety/depression.
Diagnostic Test: EuroQol Visual Analogue Scale (EQ-VAS) — records the patient's self-rated health on a vertical visual analogue scale where endpoints are labelled: 0 "best imaginable health" - 100 "worst imaginable health"

SUMMARY:
Intensive Care Units (ICU) stabilize and maintain vital functions in critically ill patients, optimizing their survival. However, patients with prolonged stays may develop Post-ICU syndrome , characterized by physical, cognitive and psychological dysfunctions. This syndrome considerably affects the quality of life of patients. The risk of post-ICU syndrome is associated with factors such as advanced age, delirium, prolonged sedation and mechanical ventilation.

The main objective of this study is to assess the temporal evolution of post-ICU syndrome in patients who required mechanical ventilation for more than 48 hours, analyzing its incidence, associated risk factors and the impact on their long-term quality of life.

This cross-sectional study evaluates the presence of post-ICU syndrome in 2025 in patients who have been admitted to the ICU during 2021 and 2024 who required invasive mechanical ventilation for more than 48 hours. Of this total, deceased persons, those who did not give their consent, and minors will not be included.

DETAILED DESCRIPTION:
Advances in intensive care have improved short-term survival rates, but survivors of prolonged ICU stays may face medium- and long-term morbidities, influenced by both the critical illness and the ICU environment. This highlights the importance of a comprehensive approach to their care, focused on improving post-ICU quality of life.

Post-intensive care syndrome is defined as the appearance or worsening of physical, cognitive and/or mental health impairments in patients who survive a stay in an ICU. This syndrome usually manifests during the first 48 hours after admission or after discharge, persisting in the long term and negatively affecting quality of life and daily functionality. In the physical field, is characterized by acquired neuromuscular weakness that frequently limits the patient's autonomy. Regarding psychological dysfunction, disorders such as anxiety, depression and post-traumatic stress disorder are observed; in the neurocognitive field, dysfunctions in memory, attention and executive functions affect daily life. This syndrome considerably affects the quality of life of patients. The risk of post-ICU syndrome is associated with factors such as advanced age, delirium, prolonged sedation and mechanical ventilation.

The main objective of this study is to assess the temporal evolution of post-ICU syndrome in patients who required mechanical ventilation for more than 48 hours.

Specific objectives:

* To establish the incidence of PICUS in patients admitted to the ICU for respiratory failure between January 2021 and December 2024.
* To identify the risk factors associated with the development of post-ICU syndrome in these patients, considering both clinical and sociodemographic factors.
* To evaluate the impact of post-ICU syndrome on the quality of life of patients over time, studying the physical, cognitive and psychological consequences of the syndrome.
* To explore the impact on their families, analyzing the emotional impact and the quality of life of caregivers.

This is a cross-sectional study, in which no experimental intervention will be carried out on the patients.

The study population will be patients hospitalized in the Intensive Care Unit between January 2021 and December 2024 undergoing mechanical ventilation for more than 48 hours. Deceased persons, those who did not give their consent, and minors will not be included. The final sample size is expected to be representative for the purposes of the study.

Data collection will be carried out through interviews in 2025, which will allow obtaining detailed information on the current situation of these patients about the presence of symptoms as a consequence of their stay in the ICU more than two years ago.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the ICU between January 2021 and December 2023 who have required invasive mechanical ventilation for a period of more than 48 hours.
* Patients who give their informed consent to participate in the study.
* Patients aged 18 years or older

Exclusion Criteria:

* Patients who have been subjected to mechanical ventilation for less than 48 hours during their stay in the ICU between January 2021 and December 2023.
* Patients who do not give their informed consent and, therefore, do not agree to participate in the interview.
* Patients who have died during their stay in the ICU or in the period between 2021 and 2024.
* Patients under 18 years of age.
* Patients in whom it is not possible to collect all the information necessary to adequately assess post-ICU syndrome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized in the ICU between January 2021 and December 2023 undergoing mechanical ventilation for more than 48 hours
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Post-Intensive Care Unit Symptoms | More than 1 year after intensive care unit discharge
  Rate of patients currently suffering of post-intensive care symptoms

SECONDARY OUTCOMES:
Quality of life assessment | More than 1 year after intensive care unit discharge
  patient's self-rated health on a vertical visual analogue scale where endpoints are labelled: 0 "best imaginable health" - 100 "worst imaginable health"

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario de Gran Canaria Doctor Negrín, Las Palmas de Gran Canaria, Las Palmas, Spain

IPD SHARING:
Plan to Share IPD: Undecided